CLINICAL TRIAL: NCT03334136
Title: The Effect of Vitamin D Supplementation on Psoriasis Severity Measured by Psoriasis Area Severity Index (PASI) in Patients With Lower Range Serum 25-hydroxyvitamin D Levels
Brief Title: The Effect of Vitamin D Supplementation on Psoriasis Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); University of Tromso (Other); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TromsøPsoriasis-2016-1; 2016-003378-42 (EudraCT Number); 2016/1789 (Other: The Regional Ethics Committee)
Record Dates: First submitted 2017-10-05; First posted 2017-11-07 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Psoriasis; Vitamin D Deficiency
MeSH Terms: conditions — Psoriasis; Vitamin D Deficiency | interventions — 25-hydroxyvitamin D

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to high dose vitamin D (20.000 IU/week) versus placebo for 4 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Active Comparator): 25-hydroxyvitamin D 20.000 IU capsule given orally. Five capsules the first day and thereafter one capsule every week for 4 months.
  Interventions: Drug: 25-Hydroxyvitamin D
- Placebo (Placebo Comparator): Placebo oral capsules. Five capsules the first day and thereafter one capsule every week for 4 months.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: 25-Hydroxyvitamin D — Capsules containing 20 000 IU 25-hydroxyvitamin D given orally: five capsules the first day and thereafter one capsule every week for 4 months (average daily dose approximately 3.000 IU)
  Other Names: Dekristol
  Arms: Vitamin D
Drug: Placebo oral capsule — Five capsules the first day and thereafter one capsule every week for 4 months.
  Arms: Placebo

SUMMARY:
The study evaluates the effect of oral vitamin D supplementation on the severity of psoriasis measured by Psoriasis Area Severity Index (PASI) in adults with lower vitamin D levels. Half of the participants will receive vitamin D, while the other half receive placebo.

DETAILED DESCRIPTION:
Studies have indicated an association between lower levels of vitamin D and increased risk of psoriasis. This study investigate if vitamin D supplementation can reduce the severity of the skin disease as measured by Psoriasis Area Severity Index (PASI), as well as positively influence the cardiometabolic profile and skin microbiota of persons with psoriasis through a winter season.

Consenting participants will be randomized to high dose vitamin D (20.000 IU/week) versus placebo for four months. The participants will be recruited based on their 25-hydroxyvitamin D (25(OH)D)-measurements in the 7th survey in the Tromsø study where 21.083 subjects attended.

In order to assure sufficient study participation we will (in season 2, winter 2018/19) include 20-40 persons from the general population in Tromsø aged 20-79, who did not partake in Tromsø 7, through advertisement and contact with patient organizations.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis diagnosis confirmed by a dermatologist at visit 1.
* Psoriasis Area Severity Index (PASI) score > 0 at inclusion.
* Serum 25 hydroxyvitamin D levels < 60 nmol/L confirmed at visit 1
* Do not meet exclusion criteria

Exclusion Criteria:

* age above 79 years
* subjects allergic to nuts (the study capsules contain peanut oil)
* subjects with primary hyperparathyroidism
* granulomatous diseases (sarcoidosis, tuberculosis, granulomatosis with polyangiitis (Wegners))
* reduced kidney function (creatinine > 130 μmol/L in males and 120 μmol/L in females)
* measured systolic blood pressure (BP) > 174 mmHg, diastolic BP > 104 mmHg
* poorly controlled diabetes (HbA1c > 9.0 %)
* renal stones the last five years
* subjects who use solarium on a regular basis (more than twice a month on average), nor can this be performed under the course of the study
* subjects who plan holiday(s) in tropical areas including the Canary Islands for more than two weeks under the course of the study
* subjects with clinical signs of proximal myopathy (problems with standing up from chair or walking stairs)
* subjects seriously physically or mentally ill and unfit for participation in a clinical study (as judged by one of the study doctors)
* subjects who have been diagnosed with or treated for organ cancer within the past 12 months (basal cell carcinoma and other limited nonmelanoma skin cancer or melanoma in situ can be included).
* pregnancy. Females of child bearing potential (below the age of 50) may participate if they use highly effective anticonception (hormonal, intrauterine device(IUD), in accordance with Clinical Trial Facilitation Group(CTFG) guidelines); if living in a relation with a partner who has been sterilized; if living in a lesbian relationship; or do not have or wish to have a male partner. If, in spite of the above, a pregnancy occurs during the study, it will lead to exclusion form the study. In females < 50 years a pregnancy test will be performed at inclusion
* subjects using vitamin D supplementation (incl. cod liver oil) above 800 IU (20 microgram) (5 ml codliver oil = 400 IU) or active vitamin D drugs (Rocaltrol or Etalpha) within the last month before study start are excluded. Furthermore, vitamin D supplements (e.g. codliver oil) or drugs apart from the study medication can not be used during the course of the study.
* subjects who during the last month before inclusion have used phototherapy/light therapy or heliotherapy as prescribed by a dermatologist, nor can this treatment be performed under the course of the study
* subjects who have started treatment with a new oral or injection drug for psoriasis or psoriasis arthritis (E.g. Methotrexate, Cyclosporine, Acitretin or biological treatment like Humira, Remicade, Stelara and others ) within the last 2 months (evaluated by dermatologist). Nor can a new oral or injection drug which influences psoriasis severity be introduced during the study. In this case the participant will be withdrawn from the study.
* subjects who have participated (been randomized) in the pilot study
* In season 1: subjects who have participated (been randomized) in the D-COR study.

Topical treatments containing vitamin D or vitamin D analogs (including Daivobet) cannot be used during the study. If a subject uses these products regularly, replacement products which only contain local steroids will be prescribed as alternates or the participant is excluded.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index (PASI) score | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in psoriasis severity measured by PASI score. Score range from 0-72, where a higher value indicates a more severe disease.

SECONDARY OUTCOMES:
Physician Global Assessment (PGA) score | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in psoriasis severity measured by PGA score.
Dermatology Quality of Life Index (DLQI) score | Baseline, 8 weeks and 4 months
  The difference in change between the vitamin D and placebo group in self-reported quality of life measured by DLQI score. Score range from 0-30 (0-1 = no effect at all on patient's life; 2-5 = small effect on patient's life; 6-10 = moderate effect on patient's life; 11-20 = very large effect on patient's life; 21-30 = extremely large effect on patient's life).
Self-administered psoriasis area and severity index (SAPASI) score | Baseline, 8 weeks and 4 months
  The difference in change between the vitamin D and placebo group in self-reported psoriasis severity measured by SAPASI score. Score range from 0-72, where a higher value indicates a more severe disease.
Use of psoriasis related medication: topical treatment I | Baseline and 4 months
  Difference in use of topical treatment measured in grams measured by type (steroid group 1-4) and amount (in milligram) between individuals in the vitamin D and placebo group. Participants will be asked to bring their current topical medication to the first appointment and the medication will be registered and weighed in grams. They will be asked to save any tube of medication which is used during the duration of the study and bring this back for the last visit. Use of medication will be used as a proxy for severity and statistical adjustment variable.
Use of psoriasis related medication: topical treatment II | Baseline, 8 weeks and 4 months
  Difference in use of topical medication measured by the type of topical treatment (steroid group 1-4) and amount of prescriptions given between individuals in the vitamin D and placebo group. Data will be collected through self-report and data on number of prescriptions given from Norwegian Prescription database by ATC code. Use of medication will be used as a proxy for severity and statistical adjustment variable.
Long term use of psoriasis related medication | 1-2 years before inclusion to 1-2 years after study end
  Difference between use of topical and/or systemic psoriasis related medication, measured through type and number of psoriasis relevant prescriptions given (data from Norwegian Prescription database by ATC code) between individuals in the vitamin D and placebo group.
Use of psoriasis related medication: systemic treatment | Baseline, 8 weeks and 4 months
  Difference in use of systemic psoriasis medication between individuals in the Vitamin D and placebo group. Data will be collected through self-report and data on number of prescriptions given from Norwegian Prescription database by ATC code. Use of medication will be used as a proxy for severity and statistical adjustment variable.
Skin microbiome | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in skin microbiome measured by 16s rRNA sequencing also compared with skin microbiome of participants with low serum vitamin D, but without psoriasis.
Immune response in serum and the skin | Baseline and 4 months
  The investigators wish to measure changes in immune response including use of inflammatory/metabolomic markers using serum and skin biopsies (healthy and plaque skin) between the study arms (placebo versus intervention with vitamin D) before and after intervention. Details concerning chosen study panel and methods will be decided in detail later based on study findings.
Genetic expression in full blood and the skin | Baseline and 4 months
  The investigators wish to measure changes in genetic expression including possible transcriptomic and proteomic analyses using full blood and skin biopsies (healthy and plaque skin) between the study arms (placebo versus intervention with vitamin D) before and after intervention. Details concerning methods will be decided in detail later based on study findings.
Cardiometabolic marker: blood pressure | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in blood pressure(BP) in mmHg. Both systolic BP and diastolic BP will be measured. Lower values are considered to be a better outcome.
Cardiometabolic marker: HbA1c | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in HbA1c in %. Lower value are considered to be a better outcome.
Cardiometabolic marker: lipids | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in lipids(total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides) in mmol/L. Lower values of total cholesterol, LDL-cholesterol and triglycerides, and higher value of HDL-cholesterol, are considered to be a better outcome.
Cardiometabolic marker: weight | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in weight in kg. Lower values are considered to be a better outcome.
Cardiometabolic marker: Body mass index (BMI) | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in body mass index (weight/ height*height; kg/m2). Lower values are considered to be a better outcome.
Cardiometabolic marker: waist circumference | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in waist circumference in cm. Lower values are considered to be a better outcome
Cardiometabolic marker: hip circumference | Baseline and 4 months
  The difference in change between the vitamin D and placebo group in hip circumference in cm. Lower values are considered to be a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Danielsen, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Jenssen M, Furberg AS, Jorde R, Wilsgaard T, Danielsen K. Effect of Vitamin D Supplementation on Psoriasis Severity in Patients With Lower-Range Serum 25-Hydroxyvitamin D Levels: A Randomized Clinical Trial. JAMA Dermatol. 2023 May 1;159(5):518-525. doi: 10.1001/jamadermatol.2023.0357. PMID 36988936